CLINICAL TRIAL: NCT00742664
Title: Behavioral Treatment of Obsessive-Compulsive Symptoms in Youth With Prader-Willi Syndrome: A Pilot Project
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Eric Storch, Ph.D., Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPWR-CBT-001
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-07

CONDITIONS: Prader Willi Syndrome; Obsessive-compulsive Disorder
Keywords: Prader-Willi Syndrome; Compulsive behavior; Hoarding; Obsessive-compulsive disorder; Children; Treatment; genetically; confirmed; diagnosis
MeSH Terms: conditions — Prader-Willi Syndrome; Obsessive-Compulsive Disorder; Compulsive Behavior; Hoarding; Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Will receive 12 sessions of twice weekly psychotherapy targeting obsessive-compulsive symptoms.
  Interventions: Behavioral: Cognitive-behavioral therapy
- 2 (Placebo Comparator)
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — The manual is informed by behavioral principles and provides a structured, replicable manner of treating OC symptoms in youth with PWS. The treatment is individual in nature, includes a strong family component (i.e., teaching parents to be their child's coach/therapist), and lasts for approximately 12 sessions, held in a twice-weekly format. In addition, the protocol includes several specific components: education about OC symptoms (i.e., etiology, behavioral function, etc.), developing a hierarchy of rituals to target, exposure and response prevention exercises, promoting adaptive familial responses to child behaviors, and relapse prevention and problem solving future situations.
  Arms: 1
Behavioral: Wait-list control — The subject will not receive active treatment during this interval.
  Arms: 2

SUMMARY:
Obsessive-compulsive (OC) symptoms are often present among youth with Prader-Willi Syndrome (PWS). They are also associated with considerable problems in the daily functioning of the child and his/her family. Although medication and behavioral treatments exist that target OC symptoms among youth without PWS, these treatments have not been thoroughly adapted for this population nor scientifically tested. Although medication has been helpful in addressing OC symptoms in several published case reports, the associated efficacy is modest and the potential for side effects is a realistic concern. Given that behavioral treatment for OC symptoms has superior efficacy to pharmacotherapy in youth without PWS without the accompanying risk for adverse side effects, it follows that an adapted version of behavioral therapy may hold promise in treating clinically problematic OC symptoms in youth with PWS. Thus, the purpose of the proposed grant is to develop and pilot-test a behavioral treatment for OC symptoms for use in youth with PWS. This study will allow us to develop and test a treatment protocol aimed at reducing OC symptoms that are clinically problematic and negatively impact functioning and quality of life in the child and his/her family.

DETAILED DESCRIPTION:
Background: Obsessive-compulsive (OC) symptoms in youth with Prader-Willi Syndrome (PWS) are commonly present and associated with considerable functional impairment to the child and his/her family. Although pharmacological and behavioral treatments exist that target OC symptoms among youth without PWS, these treatments have not been systematically adapted for this population nor rigorously tested. Furthermore, although pharmacological interventions have shown promise in PWS in case reports, the efficacy is modest and the potential for side effects has been documented in youth with and without PWS. Given that behavioral treatment for OC symptoms has superior efficacy to pharmacotherapy in youth without PWS, without the accompanying risk for adverse side effects, it follows that an adapted version of this modality may hold promise in treating clinically problematic OC symptoms in youth with PWS.

Objectives: There are two primary study objectives: First, to develop a well-specified behaviorally oriented psychotherapy protocol that addresses OC symptoms, both food and non-food related, in youth with PWS. Second, to conduct a randomized wait-list controlled trial of the protocol in 12 youth with PWS.

Study Design: There will be two phases to this study: Phase I - Therapy development/manual writing and a small open trial; and Phase II - a small wait-list controlled pilot trial. Briefly, Phase I will concentrate on developing the treatment protocol through a process that draws on expert opinion coupled with focused interviews with parents. Based on this, a preliminary manual developed by the investigators will be piloted in 6 youth with PWS. Phase II will involve a preliminary test of the protocol in a sample of 12 families. This trial will focus primarily on feasibility issues (versus efficacy) in order to refine the manual, develop process measures to evaluate therapist's competence and adherence to manualized guidelines, train evaluators in assessment tasks, and develop data collection and coding systems. Six youth will be randomized to receive the treatment protocol, while 6 will participate in a wait-list of an equivalent time period. Diagnostic and symptom severity assessments will be conducted at appropriate time points (e.g., Screening, Baseline, Post-treatment) by a blinded, trained independent evaluator.

ELIGIBILITY:
Inclusion Criteria:

1. The child must have a genetically confirmed diagnosis of PWS;
2. CY-BOCS Compulsion Score ≥ 8. The Compulsion Scale Score is being used as youth with PWS may have difficulty understanding or identifying the connection between obsessional thoughts and subsequent rituals. Therefore, use of the Total Score may provide an inaccurate depiction of symptoms (Storch et al., 2005);
3. Stable on any psychotropic medications for 8 weeks prior to study entry;
4. Between the ages of 6 and 17 years as the present measures are valid for use in this age span;
5. At least one parent available to accompany the child to all sessions; and
6. English speaking.

Exclusion Criteria:

1. Current suicidal intent or risk;
2. A positive diagnosis in the caregiver of mental retardation, psychosis, or other psychiatric conditions that would limit their ability to understand psychotherapy.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS; Scahill et al., 1997). | Baseline, Mid-Treatment, Post-treatment

SECONDARY OUTCOMES:
Clinical Global Improvement (CGI; Guy, 1976). | Mid- and Post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- All Children's Hospital, St. Petersburg, Florida, United States